CLINICAL TRIAL: NCT05137457
Title: Evaluating the Effectiveness of Cognitive Behavioral Therapy for Insomnia on Patient Centered Outcomes Such as Self Efficacy, Pain Control and Overall Quality of Life in the Young Adult Chronic Pain Population: The Young Adult CBTi (YAC)
Brief Title: Effectiveness of Cognitive Behavioral Therapy for Insomnia in Young Adults With Chronic Pain
Acronym: YAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: An RCT was not valid anymore as app has become open source and will risk a contamination of study population
Sponsor: Women's College Hospital (Other)
Collaborators: Toronto Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2020-0103-B
Record Dates: First submitted 2021-03-08; First posted 2021-11-30 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Insomnia; Chronic Pain; Insomnia Due to Medical Condition
Keywords: Insomnia; Pain
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Chronic Pain; Pain | interventions — Amyloid

STUDY DESIGN:
Intervention Model Description: Prospective pilot study with participants randomized to either the intervention Delivering Online "ZZZ's with Empirical support- DOZE app with Sleep diary/Cognitive Behavioral Therapy for insomnia- CBTi) or attention control DOZE app with Sleep diary only groups. Participants will input entries into their sleep diary as an attention control over a 10-week period. For the intervention arm, mobile CBTi will be offered using the DOZE app, an integrated smart phone app and web based self-management program. The intervention will be delivered on restricted password-protected applications that will allow adherence to be tracked. Participants will log onto the sleep dairy once a day over 10-weeks to complete sleep diary entries, develop and track their goals, and receive sleep health education tailored sleep health interventions. After 10-weeks, participants will complete questionnaires on sleep health, pain, and Health Related Quality of Life.
  Actigraphy use will be optional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following consent, participants will be randomized and allocated to either the intervention or control arm of the trial. Randomization will be centrally controlled, and allocation will be concealed using a secure, web-based randomization on the Research Electronic Data Capture (REDCap) platform. The patients, the clinical care team (pain physicians, sleep physician, occupational therapist, and social worker), outcome adjudicators and the study statisticians will all remain blinded to randomization and group allocation. The personnel teaching the app to the intervention group will be aware of group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delivering Online "ZZZ's with Empirical support (DOZE) app (Experimental): The mobile Cognitive Behavioral Therapy for insomnia (CBTi) will be offered using the Delivering Online "ZZZ's with Empirical support (DOZE) app. Patients assigned to the intervention group will be given the DOZE app which is an integrated smart phone app and web based self-management program for adolescents and young adults with sleep problems. The intervention will be delivered on restricted password-protected application. Participants will be encouraged to log onto the sleep dairy once a day over 10-weeks to complete sleep diary, develop and track their goals, and receive sleep health education tailored sleep health interventions. After 10-weeks, participants will complete questionnaires on sleep health, pain, and Health Related Quality of Life (HQRL). The use of actigraphy will be optional in view of the COVID19 pandemic.
  Interventions: Other: Delivering Online "ZZZ's with Empirical support (DOZE) app; Other: Sleep diary
- Sleep Diary Only Attention Control (Active Comparator): The control group will receive the control version of the DOZE app where the patients will be able to access the sleep diary only, without the CBTi intervention. Participants will simply use the app to input entries into their sleep diary as an attention control over a 10-week period.
  After the 10-week intervention period, participants will again complete a battery of questionnaires on sleep health, pain, and HRQL. The use of actigraphy will be optional in view of the COVID19 pandemic.
  Interventions: Other: Sleep diary

INTERVENTIONS:
Other: Delivering Online "ZZZ's with Empirical support (DOZE) app — The DOZE app is a unique digital CBTi intervention that can be used on any mobile phone, tablet or computer, using the iPhone Operating System (iOS) or Android software. It is an innovative program that consists of an integrated smart phone app and web self-management system ("DOZE") to help adolescents and young adults to sleep better. It allows data capture through entries in a sleep diary and calculation of specific clinical indices. The acquisition of baseline sleep health data over a two-week period is then used to provide personalized targets and tailored therapeutic interventions during the treatment phase. The app also includes a self-monitoring tool that fosters goal setting and provides feedback on sleep and goal attainment. DOZE allows for real time assessment of sleep related behaviors and customized reports and graphs from the young adults' data. The app provides reminders about specific goals and positive feedback (increasing scores) for each step towards a goal.
  Arms: Delivering Online "ZZZ's with Empirical support (DOZE) app
Other: Sleep diary — The control group will receive the control version of the DOZE app where the patients will be able to access the sleep diary only, without the CBTi intervention. Participants will simply use the app to input entries into their sleep diary as an attention control over a 10-week period.

SUMMARY:
The aim of the Young Adult Cognitive Behavioral Therapy (YAC) study is to evaluate the effectiveness of the Delivering Online "ZZZ's with Empirical support (DOZE) app, a unique digital cognitive behavioral therapy for insomnia (CBTi) in young adult patients with chronic pain.

DETAILED DESCRIPTION:
Sleep, activity, and pain interactions have the potential to impact almost all important protective and regulatory processes in the body. Long-term sleep disruption is associated with increased pain sensitivity, prolonged pain duration, and development of chronic pain. Degree of pain relief can directly impact the quality and disruption of sleep, mood, behavior, social participation, and has a devastating impact on Health Related Quality of Life (HRQL).

Cognitive behavioral therapy for insomnia (CBTi) is a behavioral modification approach and is currently a frontline therapy for adults with sleep disorders. However, CBTi is still in early stages of development for adolescent and young adult populations, and less so for youth with comorbid mental and physical health conditions and chronic pain.

Primary aim: Assess the feasibility of implementing the DOZE app.

Secondary aim: 1). To examine the variance in effectiveness outcomes, including sleep health, pain, and overall Health Related Quality of Life (HRQL). 2). To determine the required sample size for a future definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Young adult patients aged 18 - 25 years old, who have
* Non-malignant chronic pain lasting more than 3 months, with
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for insomnia,
* English speaking with
* Access to a mobile phone or a computer with internet access.

Exclusion Criteria:

* Patients who require urgent CBT treatment as per their health care provider
* Patients who have received CBT in the past 3 months
* Patients participating in other psychological treatments and/or drug trials during the study
* Patients who have other significant medical conditions- Life threatening (e.g. cancer), neurological conditions (e.g. epilepsy)
* Patients who have other significant psychiatric conditions-Severe depression or active suicide intent
* Situations resulting in forced sleep disruption or derangement of sleep schedule such as night shift work > 2 nights per week in the past 3months, pregnancy or breastfeeding.
* Inability to communicate with health care providers or the research personnel
* Inability to fill out self-report questionnaires, study materials, or follow instructions.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Study recruitment/retention | 1 year
  Number of Participants recruited/dropping out of study (accrual/dropout rates)
Study compliance to DOZE app intervention/Sleep diary | 10 weeks
  Number of Participants completing/using the DOZE app and completing the sleep diary during 10 weeks study intervention
Study DOZE app treatment evaluation | 12 weeks
  Participants' scoring on a 5 point Likert scale pre and post study intervention

SECONDARY OUTCOMES:
Patient reported improvement in sleep & pain | 12 weeks
  Number of Participants reporting Pain Inventory & Sleep Health improvement on a scale of 0 to 10
Patient reported improvement in Health Related Quality Of Life | 12 weeks
  Number of Participants reporting an improvement in HRQOL in Questionnaire
Patient reported Global Impression of Change | 12 weeks
  Number of Participants reporting an improvement in PGIC in Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada